# **Replication of the LEAD-2 Trial in Healthcare Claims**

**RCT DUPLICATE – LEAD-2** 

August 4, 2021

#### 1. RCT Details

This section provides a high-level overview of a **published** RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Efficacy and Safety Comparison of Liraglutide, Glimepiride, and Placebo, All in Combination With Metformin, in Type 2 Diabetes. The LEAD (Liraglutide Effect and Action in Diabetes)-2 study (NCT00318461).

#### 1.2 <u>Intended aim(s)</u>

To assess whether the glycemic control achieved by adding liraglutide to metformin was non-inferior to glimepiride and metformin combination therapy after 26 weeks of treatment, in subjects with type 2 diabetes and previously treated with oral antidiabetic therapy.

#### 1.3 Primary endpoint for replication

Long-term glycemic control defined as change in HbA1c from baseline to the end of follow-up.

## 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

The sample size calculation was based on both HbA1c and body weight endpoints. The assumed standard deviation for HbA1c and the coefficient of variance for body weight were 1.2% and 3%, respectively. The combined power (calculated as the product of the marginal powers for HbA1c and body weight) was at least 85%. Noninferiority of glycemic control with liraglutide versus glimepiride was concluded if the upper limit of the two-sided 95% CI for the treatment difference was < 0.4%.

With a standard deviation of 1.2% for HbA1c and a coefficient of variance of 3% for body weight, it was concluded that at least 168 subjects were required to complete the treatment in the liraglutide and in the glimepiride, respectively. Assuming a dropout rate of 25% after 26 weeks of treatment, the number of subjects to be randomized was calculated to be 228 in each of the liraglutide and glimepiride treatment groups.

# 1.5 <u>Secondary endpoint for replication (assay sensitivity) and RCT finding</u> n/a

#### 1.6 Trial estimate

The HbA1c mean decreases of 1.0% ( $\pm$  0.1) for both the 1.2 and 1.8 mg/day liraglutide groups and 1.0% ( $\pm$  0.1) for glimepiride group. Treatment difference in HbA1c was 0.0% [95% CI: -0.2 to 0.2] for both comparisons liraglutide 1.2 mg/day versus glimepiride and liraglutide 1.8 mg/day versus glimepiride (Nauck M et al. 2009).

### 2. Person responsible for implementation of replication in Aetion

Elvira D'Andrea, MD, MPH, implemented the study design in the Aetion Evidence Platform and SAS 9.4. She is not responsible for the validity of the design and analytic choices. All implementation steps are recorded, and the implementation history is archived in the platform.

## 3. Data Source(s)

Optum CDM

## 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

Figure 1. Design Diagram - LEAD-2 TRIAL REPLICATION



#### 5. Cohort Identification

#### 5.1 Cohort Summary

This study will involve a new user, parallel group, propensity score-matched, retrospective cohort design comparing injectable subcutaneous liraglutide (1.2 or 1.8 mg/day) to oral glimepiride (4 mg once daily). Treatments in both arms are administered in combination with metformin (up to 2,000 mg/day). Patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of liraglutide or glimepiride. The analyses will be restricted to individuals with type 2 diabetes mellitus who have been previously treated with antidiabetic drugs. In the replication, previous anti-diabetic treatment was defined as the presence of at least 2 prescriptions for metformin within 6 months before and including cohort entry.

#### 5.2 Important steps for cohort formation

New use of liraglutide (exposure) is defined as no use of the exposure drug within 180 days prior to index date. New use of glimepiride (comparator) is defined as no use of the comparator drug within 180 days prior to index date. Eligible patients are required to be new users with respect to both exposure and comparator groups (i.e., no use of both exposure and comparator drugs) within 180 days prior to index date.

#### 5.2.1 Eligible cohort entry dates

Liraglutide indication as an adjunct to diet and exercise to improve glycemic control in adults with type 2 diabetes mellitus was approved by FDA on Jan 25, 2010 (the approval of glimepiride for the same indication was antecedent to 2010). Thus, the initial eligible cohort entry date is the first date after the FDA approval available in the data. The last eligible date is June 30, 2020, three months before the end of all available data in Optum CDM. Since the effects of liraglutide and glimepiride on the outcome (i.e., change in HbA1c) will be estimated between 56 and 212 days after cohort entry (see Section 6.3), this will allow all eligible patients to contribute to the outcome. The database used is Optum CDM because lab results/values are available in this database for a subset of laboratory tests, including the A1C tests. The following eligible cohort entry dates were included:

- Optum CDM: Jan 26, 2010 Jun 30, 2020
- 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

<u>Note</u>. Patients who are censored between cohort entry and the beginning of the outcome assessment window (i.e., 0.x-56 days after cohort entry) for the reasons reported in the Section 6.3.2 will not contribute to the unmatched or matched cohorts. Further details on the number of patients who are excluded from the study cohort are reported in the Section 7.

## 5.3 Flowchart of the study cohort assembly

For liraglutide vs. glimepiride: Aetion link: https://bwh-dope.aetion.com/cohorts/details/23482/1688/71700

| | Optum | |
|---|---|---|
| | Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 79,335,559 |
| Did not meet cohort entry criteria | -78,554,666 (99%) | 780,893 |
| Excluded due to insufficient enrollment | -119,528 (15%) | 661,365 |
| Excluded due to prior use of referent | -424,186 (64%) | 237,179 |
| Excluded due to prior use of exposure | -138,679 (58%) | 98,500 |
| Excluded because patient qualified in >1 exposure category | -85 (<1%) | 98,415 |
| Excluded based on nursing home admission in the prior 180 days | -3,784 (4%) | 94,631 |
| Excluded based on gender missing or unknown | -10 (<1%) | 94,621 |
| Excluded based on Inclusion #1.1 - Type 2 diabetes mellitus | -6,027 (6%) | 88,594 |
| Excluded based on Inclusion #1.2 - Metformin use (2 prescriptions within 183 days) | -55,832 (63%) | 32,762 |
| Excluded based on Inclusion #1.3 - Concomitant initiation or concurrent use of metformin | -3,670 (11%) | 29,092 |
| Excluded based on Inclusion #1.4 - No use of other anti-diabetic meds | -9,861 (34%) | 19,231 |
| Excluded based on Inclusion #2.1 - 3 records of HbA1c 2-20% values/results within 365 days | -13,962 (73%) | 5,269 |
| Excluded based on Inclusion #2.2 - At least 1 lab value HbA1c 7-11% recorded within 90 days | -808 (15%) | 4,461 |
| Excluded based on Inclusion #3.1 - Age > 18 | -0 (<1%) | 4,461 |
| Excluded based on Inclusion #3.2 - Age < 80 | -87 (2%) | 4,374 |
| Excluded based on Exclusion #1 - Morbid Obesity BMI > 40 | -147 (3%) | 4,227 |
| Excluded based on Exclusion #2 - Any insulin use | -234 (6%) | 3,993 |
| Excluded based on Exclusion #3 - End-stage liver disease | -9 (<1%) | 3,984 |
| Excluded based on Exclusion #4 - Viral Hepatitis B and C | -7 (<1%) | 3,977 |
| Excluded based on Exclusion #5 - CKD stage 5, End-stage renal disease, dialysis, or renal transplant | -0 (<1%) | 3,977 |

| Excluded based on Exclusion #6.1 - Myocardial Infarction | -1 (<1%) | 3,976 |
|---|---|---|
| Excluded based on Exclusion #6.2 - Heart Failure | -1 (<1%) | 3,975 |
| Excluded based on Exclusion #7 - Anti-VEGFi OR Photocoagulation | -5 (<1%) | 3,970 |
| Excluded based on Exclusion #8 - Uncontrolled hypertension | -34 (<1%) | 3,936 |
| Excluded based on Exclusion #9 - Malignant neoplasm (except non-melanoma skin cancer) | -79 (2%) | 3,857 |
| Excluded based on Exclusion #10 - Recurrent Hypoglycemia | -8 (<1%) | 3,849 |
| Excluded based on Exclusion #11 - Systemic glucocorticoids use | -48 (1%) | 3,801 |
| Excluded based on Exclusion #12 - Drug addiction or alcohol abuse and dependence | -11 (<1%) | 3,790 |
| Excluded based on Exclusion #13 - Mental incapacity, unwillingness to comply | -13 (<1%) | 3,777 |
| Excluded based on Exclusion #14 - Pregnancy | -0 (<1%) | 3,777 |
| Excluded based on Exclusion #15.1 - Type 1 diabetes mellitus (contraindication glimepiride) | -10 (<1%) | 3,767 |
| Excluded based on Exclusion #15.2 - Diabetic ketoacidosis (contraindication glimepiride) | -2 (<1%) | 3,765 |
| Excluded based on Exclusion #15.3 - Other metabolic acidosis (contraindication glimepiride) | -1 (<1%) | 3,764 |
| Excluded based on Exclusion #16 - Multiple endocrine neoplasia type 2 (MEN2) | -0 (<1%) | 3,764 |
| Final cohort | | 3,764 |

#### 6. Variables

## 6.1 Exposure-related variables:

### Study drug:

New initiation of injectable subcutaneous liraglutide (1.2 or 1.8 mg/day), a glucagon-like peptide-1 receptor agonist. New initiation is defined as no use of liraglutide within 180 days before treatment initiation (washout period). New users of liraglutide are not allowed to receive glimepiride within 180 days prior to treatment initiation. Concurrent use of metformin is required (2,000 mg/day).

## Comparator agent:

New initiation of oral glimepiride (4 mg once daily). New initiation is defined as no use of glimepiride within 180 days before treatment initiation (washout period). New users of glimepiride are not allowed to receive liraglutide within 180 days prior to treatment initiation. Concurrent use of metformin is required (2,000 mg/day).

#### 6.2 Preliminary Covariates:

- Age
- Gender
- Combined Comorbidity Index (CCI), measured over the baseline covariate assessment period, defined as 180 days prior to and including index date.

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (Appendix B).

### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcome variables of interest (definitions provided in **Appendix A**):

• **Primary outcome:** Changes in HbA1c from baseline to 26 weeks of treatment (end of follow-up).

Note. In the trial, HbA1c was also measured at 8, 12, 18 weeks (± 3 days) after randomization. Missing values of HbA1c at 26 weeks were replaced using last observation carried forward (LOCF) in the intention-to-treat (ITT) analysis set. In the replication, HbA1c at baseline will be defined as the last recorded HbA1c value measured within 90 days before and including cohort entry date in both groups. HbA1c at the end of follow-up will be defined as a recorded HbA1c value closest to the end of the 26<sup>th</sup> week and measured between 56 and 212 days (8-30 weeks) after cohort entry.

Secondary outcome: --

### 6.3.2 Primary analysis and study follow-up

As-treated (AT) analysis will be performed as main analysis. The treatment drug will be defined as the index drug assigned on the day of cohort entry. Patients will be followed for about 30 weeks (212 days). Compared to the trial (Nauck M et al. 2009), we will

extend the follow-up and the outcome assessment periods of 4 weeks. The follow-up and outcome assessment window will start 56 days after cohort entry date and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest (measured between 56 and 212 days after cohort entry),
- The date of end of continuous registration in the database (disenrollment or end of available data),
- End of the study period,
- Measured death event occurs,
- Index drugs discontinuation (liraglutide, glimepiride or metformin),
- Crossover or addition of drug from the other treatment group,
- Addition of any other anti-diabetic medications,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.

<u>Note</u>. To decrease the incidence of missing values of the outcome (specifically, missing of HbA1c values measured between 56-212 days after cohort entry), we required that the eligible patients had at least 3 HbA1c measurements recorded within 365 days before and including cohort entry. This will increase the probability of including in the final cohort patients who are adherent to a routinely HbA1c testing and, consequently, will decrease the frequency of missing values of the outcome. Multiple imputation will be used to handle missing values in the primary analysis, while complete case analysis will be applied in a sensitivity analysis.

#### 7. Initial Feasibility Analysis

## Aetion report name:

For liraglutide vs. glimepiride

Optum CDM (continuous HbA1c outcome) https://bwh-dope.aetion.com/projects/details/1688/rwrs/71723

Optum CDM (binary HbA1c outcome [flag: presence or absence of an HbA1c result within 56-212 days after cohort entry]) – calculated merging the databases from  $\frac{https://bwh-dope.aetion.com/projects/details/1688/rwrs/71715}{https://bwh-dope.aetion.com/projects/details/1688/rwrs/71715}$  and  $\frac{https://bwh-dope.aetion.com/projects/details/1688/rwrs/71715}{https://bwh-dope.aetion.com/projects/details/1688/rwrs/71715}$ 

<u>dope.aetion.com/projects/details/1688/rwrs/71716</u> – see file LEAD-2\_programming\_steps and output of "STEP 1 - Initial FEASIBILITY Analysis (with study outcome) - Paragraph 7 of the protocol"

Date conducted: 06/17/2021

Complete Aetion feasibility analysis using age and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will mean and standard deviation of the HbA1c outcome stratified by treatment group.

## • Report patient characteristics by treatment group For liraglutide vs. glimepiride

| | Optum CDM | | |
|---|---|---|---|
| | Glimepiride - Comparator | Liraglutide - Exposure | Difference |
| Number of patients * | 3,096 | 378 | - (-, -) |
| Age | | | |
| mean (sd) | 64.24 (10.37) | 59.22 (10.94) | 5.02 (3.90, 6.13) |
| median [IQR] | 67.00 [58.00, 72.00] | 60.00 [51.00, 68.00] | - (-, -) |
| Gender | | | |
| M = MALE; n (%) | 1,726 (55.7%) | 179 (47.4%) | 8.39% (3.08%, 13.7%) |
| F = FEMALE; n (%) | 1,370 (44.3%) | 199 (52.6%) | -8.39% (-13.7%, -3.08%) |
| Combined Comorbidity Score - CCI (180 days) | | | |
| mean (sd) | 2.06 (1.56) | 1.86 (1.36) | 0.19 (0.03, 0.36) |
| median [IQR] | 2.00 [1.00, 3.00] | 2.00 [1.00, 2.00] | - (-, -) |

<sup>\*</sup> The overall n. of patients in the unmatched cohort is 3,470. Patients who were censored between cohort entry and the beginning of the outcome assessment window (n. 290 patients) are excluded from the Table reporting patient characteristics by groups because they will not contribute to the unmatched or matched cohorts.

# • Report summary parameters of study population **FEASIBILITY- FOR STUDY OUTCOME For** liraglutide vs. glimepiride

| | Optum CDM |
|---|---|
| Number of patients in full cohort | 3,764 |
| Number of patients that did not begin follow-up * | 290 |
| Number of patients | 3,474 |
| Number of person-years of patients that did begin the follow-up | 1,118.53 |
| Number of patients in group: Glimepiride | 3,096 |
| Number of patients in group: Liraglutide | 378 |
| Outcome - Lab value HbA1c | |
| mean (sd) | 7.24 (1.01) |
| median [IQR] | 7.00 [6.60, 7.70] |
| minimum | 4.1 |
| maximum | 13.4 |
| Number of patients with zero value | 0 |
| Non-zero mean value (SD) | 7.24 (1.01) |
| Non-zero median value [IQR] | 7.00 [6.60, 7.70] |

<sup>\*</sup> patients who were censored between cohort entry and the beginning of the outcome assessment window/follow-up (i.e., 0.5-56 days after cohort entry) will not contribute to the unmatched and matched cohorts.

## • Report median follow-up time by treatment group For liraglutide vs. glimepiride

| Median Follow-Up Time (Days) [IQR] – AT analysis | |
|--------------------------------------------------|---------------|
| Patient Group Optum CDM | |
| Overall Patient Population | 99 [84, 148] |
| Referent | 101 [84, 148] |
| Exposure | 88 [79, 130] |

• Report reasons for censoring in the overall study population

#### • For liraglutide vs. glimepiride

| | Overall (n. 3,470) | Liraglutide (n. 378) | Glimepiride (n. 3,092) |
|---|---|---|---|
| Outcome * | 2,262 (65.2%) | 233 (61.6%) | 2,029 (65.6%) |
| Death | 2 (0.1%) | 0 (0%) | 2 (0.1%) |
| Start of an additional exposure | 8 (0.2%) | 3 (0.8%) | 5 (0.2%) |
| End of index exposure | 368 (10.6%) | 74 (19.6%) | 294 (9.5%) |
| Maximum follow-up time | 336 (9.7%) | 22 (5.8%) | 314 (10.2%) |
| End of patient data | 37 (1.0%) | 3 (0.8%) | 34 (1.1%) |
| End of patient enrollment | 108 (3.1%) | 12 (3.2%) | 96 (3.1%) |
| Start of additional antidiabetic drugs + Nursing home + Metformin discontinuation with allowed 60 days gap | 349 (10.1%) | 22 (5.82%) | 314 (10.2%) |

<sup>\*</sup> patients with outcome recorded between 56-212 days after cohort entry.

## • Report overall mean (sd) of the primary outcome.

| | Optum CDM |
|------------------------------------|-------------|
| Outcome – Lab value HbA1cmean (sd) | 7.24 (1.01) |

#### 8. Initial Power Assessment

### Analysis report name:

For liraglutide vs. glimepiride

Optum CDM – see file LEAD-2\_programming\_steps and output of "STEP 2 - INITIAL POWER Assessment - PS matching on age, gender, CCI (with dummy outcome) - Paragraphs 8 of the protocol"

Date conducted: 06/16/2021

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage.

Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, gender and combined comorbidity index. Power calculations are based on the formulas from Julios et al. (2008).

• Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.

#### o Optum CDM

| Non-inferiority Analysis | |
|--------------------------------|------|
| Standard deviation of outcome | 1.01 |
| Non-inferiority limit | 0.4 |
| Alpha (2-sided) | 0.05 |
| Power (1-beta) | 90% |
| Sample size required per group | 110 |
| Total sample size required | 220 |
| Number of patients matched | 752 |
| Reference | 376 |
| Exposed | 376 |

• Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: | 07/16/2021 |
|-------------------------|--------------|----------------|------------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 08/2/2021 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 9. Balance Assessment

For liraglutide vs. glimepiride

Optum CDM: see file LEAD-2\_programming\_steps and output of "STEP 3 - BALANCE Assessment (with dummy outcome) - Paragraphs 9-10 of the protocol"

Date conducted: 06/16/2021

After review of initial feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

• Report covariate balance after matching.

Note- For Table 1, please refer to **Appendix B**.

• Report reasons for censoring by treatment group.

| | Overall<br>(n. 746) | Liraglutide – exposure<br>(n. 373) | Glimepiride – comparator (n. 373) |
|---|---|---|---|
| Outcome (dummy) | 0 (0%) | 0 (0%) | 0 (0%) |
| Death | 0 (0%) | 0 (0%) | 0 (0%) |
| Start of an additional exposure | 9 (1.2%) | 6 (0.8%) | 3 (0.4%) |
| End of index exposure | 194 (26.0%) | 137 (18.4%) | 57 (7.6%) |
| Maximum follow-up time | 340 (45.6%) | 137 (18.4%) | 203 (27.2 %) |
| End of patient data | 5 (0.7%) | 3 (0.4%) | 2 (0.3%) |
| End of patient enrollment | 61 (6.3%) | 25 (3.4%) | 36 (4.8%) |
| Start of additional antidiabetic drugs + Nursing home + Metformin discontinuation with allowed 60 days gap | 137 (18.4%) | 65 (8.7%) | 72 (9.7%) |

• Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | | |
|---|---|---|---|
| Patient Group | Overall (n. 746) | Liraglutide (n. 373) | Glimepiride (n. 373) |
| Overall Patient Population | 188 [97 - 212] | 150 [89 - 212] | 212 [119 -212] |

• Report overall mean (sd) of the primary outcome (from initial feasibility analysis).

| | Optum CDM |
|------------------------------------|-------------|
| Outcome – Lab value HbA1cmean (sd) | 7.24 (1.01) |

#### **10. Final Power Assessment**

## Date conducted:

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.

| Non-inferiority Analysis | |
|--------------------------------|------|
| Standard deviation of outcome | 1.01 |
| Non-inferiority limit | 0.4 |
| Alpha (2-sided) | 0.05 |
| Power (1-beta) | 90% |
| Sample size required per group | 110 |
| Total sample size required | 220 |
| Number of patients matched | 746 |
| Reference | 373 |
| Exposed | 373 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: | 07/16/2021 |
|-------------------------|--------------|----------------|------------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 08/2/2021 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

## 11. Study Confidence and Concerns

Deadline for voting on study confidence and listing concerns:

Date votes and concerns are summarized:

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the success of the RWD study in the <a href="Google Form">Google Form</a>. This form also provides space for reviewers to list any concerns that they feel may

contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the individual respondent.

• After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

### 12. Register study protocol on clinicalTrials.gov

#### Date conducted:

• Register the study on <u>clinicalTrials.gov</u> and upload this document.

## 13. Comparative Analyses

Aetion report name:

Date conducted:

- 13.1 For primary analysis:
- 13.2 For sensitivity analyses:

## 14. Requested Results

## 14.1 <u>Table 1: Baseline characteristics before and after adjustment</u>

| Variable | Before adjustment | | After adjustment | | | |
|---|---|---|---|---|---|---|
| | Referent | Exposure | Std. diff. | Referent | Exposure | Std. diff. |
| Number of patients | | | - | | | - |
| Age categories | | | | | | |

## 14.2 <u>Table 2: Follow-up time</u>

| Patient Group | Median Follow-Up Time (Days) [IQR] |
|----------------------------|------------------------------------|
| Overall Patient Population | |
| Referent | |
| Exposure | |

## 14.3 <u>Table 3: Censoring events</u>

| | Overall | Referent | Exposure |
|---------------------------------|---------|----------|----------|
| Outcome | | | |
| Death | | | |
| Start of an additional exposure | | | |
| End of index exposure | | | |
| Specified date reached | | | |
| End of patient data | | | |
| End of patient enrollment | | | |

## 14.4 <u>Table 4: Results from primary analyses;</u>

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

## 14.5 <u>Table 5: Results from secondary analyses.</u>

#### 15. References

Nauck M, Frid A, Hermansen K, Shah NS, Tankova T, Mitha IH, Zdravkovic M, Düring M, Matthews DR; LEAD-2 Study Group. Efficacy and safety comparison of liraglutide, glimepiride, and placebo, all in combination with metformin, in type 2 diabetes: the LEAD (liraglutide effect and action in diabetes)-2 study. Diabetes Care. 2009 Jan;32(1):84-90. doi: 10.2337/dc08-1355.

Julious SA. Sample sizes for clinical trials with Normal data. Statist. Med. 2004; 23:1921-1986. Sealed Envelope Ltd. 2012. Power calculator for continuous outcome non-inferiority trial. [Online] Available from: https://www.sealedenvelope.com/power/continuous-noninferior/ [Accessed Fri May 07, 2021].

| # | LEAD-2 trial definitions | Implementation in routine care | | for further details or any missing information:<br>618wrywYjEaXzfLTcuK-VCenb6b-gV?usp≕sharing |
|---|---|---|---|---|
| | Trial details - clini | ICD-10 codes are not listed in this document because of excel cell size limitations and excessive number of ICD-10 codes. Full ICD-10 code lists will be available in the above Google Drive Folder (link above). ICD-9 to ICD-10 code conversions were completed using a SAS macro that implements forward/backward mapping based on the CMS ICD-9 to ICD-10 mapping: https://www.nber.org/data/icd/9-icd-10-cm-and-nex-crosswalk-general-equivalence-mapping.html | | |
| | EXPOSURI | E vs. COMPARISON | References/Rationale | Color coding |
| | Exposure: Liraglutide s.c. 0.6 mg/day, 1.2 mg/day and 1.8 mg/day in combination with metformin (1500-2000 mg/day) for 26 weeks Reference for non-inferiority: Glimepiride (4 mg/day) in combination with metformin (1500-2000 mg/day) Reference for superiority: Metformin monotherapy (1500-2000 mg/day) Aim: To evaluate whether the effect on glycaemic control (as measured by change in HbA1c) of treatment with 0.6 mg/day, 1.2 mg/day and 1.8 mg/day of liraglutide in combination with metformin was superior to metformin monotherapy and non-inferior to metformin and glimepiride combination therapy after 26 weeks of treatment. | Exposure: new-use of Liraglutide (washout 180 days) in combination with metformin NDC Generic Name: LIRAGLUTIDE NDC Brand name: Viktoza (FlexPen) Reference: new use of Glimepiride (washout 180 days) in combination with metformin NDC Generic Name: GLIMEPIRIDE NDC Brand name: GLIMEPIRIDE AMARYL | | Criteria |
| | PRIMA | RY OUTCOME | | Adequate mapping in claims |
| | Change in HbA1c from baseline to week 26 Note: in the trial missing values are replaced with last value carried forward [LVCF] | Measured as change in HbA1c from baseline to the last recorded HbA1c value between 56 and 212 days after drug initiation: <u>Loinc codes:</u> 17855-8, 17856-6, 41995-2, 43150-2, 4548-4, 4549-2, 55454-3, 71875-9, 74246-0 | | Intermediate mapping in claims |
| | INCLUS | SION CRITERIA | | Poor mapping or cannot be measured in claims |
| 0 | Informed consent obtained before any trial-related activities (trial-related activities are any procedure that would not have been performed during normal management of the subject). | N/A | | Can't be measured in claims but not important for the analysis |
| 1 | (1.1) Subjects diagnosed with type 2 diabetes and (1.2) treated with OAD(s) for at least three months. | 1.1 Selecting patients with a diagnosis of type 2 diabetes measured from the time of enrollment to the day of drug initiation inpatient (any position), outpatient (any position): Type 2 diabetes: 1.1 Selecting patients with at least two prescriptions of metformin within 183 days before cohort entry (OADs treatment ≥ 3 months), and 1.3 Concomitant or current use of metformin at cohort entry date in both treatment groups: Generic name: Metformin Hel 1.4 Selecting patients with no other anti-diabetic treatments within the 180 days before cohort entry: | | |
| 2 | HbA1c: -7.0-10.0% (both incl.) in subjects on OAD combination therapy -7.0-11.0% (both incl.) in subjects on OAD monotherapy. | 2.1 Selecting patients with 3 measurements of HbA1c values (between 2-20%) recorded within 365 days prior to and including cohort entry: Loine codes: 17855-8, 17856-6, 41995-2, 43150-2, 4548-4, 4549-2, 55454-3, 71875-9, 74246-0 AND Result value 2-20% 2.2 Selecting patients with at least one measurement of HbA1c value (between and included 7-11%) recorded within the last 91 days prior to and including cohort entry: Loine codes: 17855-8, 17856-6, 41995-2, 43150-2, 4548-4, 4549-2, 55454-3, 71875-9, 74246-0 AND Result value 7-11% | | |
| 3 | Age 18-80 years, both inclusive (as allowed according to local guidelines for metformin and glimepiride treatment). This inclusion criterion has been modified for Site 344 in Australia according to Substantial Protocol Amendment No. 1-AU, see Section 9.8.1. | Female and male, 18-80 years at the time of drug initiation | | |
| | EXCLU | | ] | |

| | | Measured 180 days prior to and including the day of drug initiation inpatient (any position), outpatient (any position): |
|---|---|---|
| 1 | Body mass index (BMI) >= 40.0 kg/m2. | Morbid obesity diagnosis or BMI >= 40 kg/m2:<br>ICD 9 diagnosis: 278.01, 278.03, V85.4x<br>ICD 10 diagnosis: E66.01, E66.2, Z68.4x |
| | | NB. Codes for bariatric surgey, complications of bariatric surgery and prescriptions of drugs for weight loss were not included in the measure since this exclusion criterion aims to exclude specifically patients with morbid obesity. Codes for obesity during pregnancy were not included because of the exclusion criterion #17. |
| | | Measured 180 days prior to and including the day of drug initiation: |
| | | NDC Generic Name: |
| 2 | Treatment with insulin within the last three months prior to trial (except for short-term treatment due to intercurrent illness at the discretion of the investigator). | Please refer to <i>Insulin</i> in "Anti-diabetic treatments" |
| | | NB. Although the trial excluded patients in treatment with insulin within the 90 days before drug initiation, with real-<br>world data we are required to be more conservative and to extend the washout period to 180 days. In fact, a 90-day<br>washout applied in real world does not garantee the exclusion of prevalent users (i.e. patients on active insulin therapy)<br>from the cohort. |
| | | Measured 180 days prior to and including the day of drug initiation in any diagnosis position and inpatient or outpatient care setting: |
| 3 | Impaired liver function, defined as alanine aminotransferase (ALAT) $\geq$ = 2.5 times upper limit of normal (one retest analysed at the central laboratory within a week is permitted with the result of the last sample being conclusive). | Cirrhosis. ICD-9 Diagnosis: 571.2, 571.5, 571.6 ICD-10 Diagnosis: K70.11, K70.2, K70.3x, K70.4x, K74.x Hepatic decompensation: |
| | | ICD-9 Diagnosis: 456.0, 456.20, 456.1, 456.21, 789.5, 789.59, 572.2, 567.0, 567.2, 567.21, 567.22, 567.29, 567.8, 567.89, 567.9, 572.4 ICD-10 Diagnosis: R18.x, 185.x, K72.x, K65.x, K66.x, K67 HCC is already excluded with exclusion criterion 9 |
| | | Measured 180 days prior to and including the day of drug initiation in any diagnosis position and inpatient or outpatient care setting: |
| 4 | Subjects known to be Hepatitis B antigen or Hepatitis C antibody positive. | Viral hepatitis B or C:<br>ICD-9 diagnosis: 070.2x, 070.3x, 070.4x, 070.51, 070.54, 070.71, 070.74, V02.61, V02.62<br>ICD-10 diagnosis: B16.x, B17.0, B17.1x, B18.0-B18.2, B19.1x, B19.2x, Z22.51, Z22.52 |
| | | Measured 180 days prior to and including the day of drug initiation in any diagnosis position and inpatient or outpatient care setting: |
| 5 | Impaired renal function defined as serum creatinine $>= 135 \mu moVL$ ( $>= 1.5 mg/dL$ ) for males and $>= 110 \mu moVL$ ( $>= 1.3 mg/dL$ ) for females (one retest analysed at the central laboratory within a week is permitted with the result of the last sample being conclusive) | CKD stage 5. End-stage renal disease, dialysis or renal transplant; ICD-9 diagnosis: 585.5, 585.6, 996.81, V42.0, V45.1x, V56.xx ICD-9 procedure: 39,95, 54.98, 55.6x ICD-10 diagnosis: N18.5, N18.6, R88.0, T82.41, T82.42, T82.49, T85.611, T85.621, T85.631, T86.1x, Y84.1, Z48.22, Z49.xx, Z91.15, Z94.0, Z99.2 ICD-10 procedure: 0TY00Zx, 0TY10Zx, 3E1M39Z, 5A1Dx0Z CPT: 50360, 50365, 90920, 90921, 90924, 90925, 90935, 90937, 90939, 90940, 90945, 90947, 90957, 90958, 90959, 90960, 90961, 90962, 90965, 90966, 90969, 90970, 90989, 90993, 90999, 9097, 99512, 99559, 99512, G0257, G0314, G0315, G0314, G0315, G0316, G0317, G0318, G0319, G0327, G0333, G0326, G0327, S0333, S0330, |
| | | Measured 180 days prior to and including the day of drug initiation in inpatient care setting, any position: |
| 6 | Clinically significant active cardiovascular disease including history of myocardial infarction within the past 6 months and/or heart failure (New York Heart Association class III and IV) at the discretion of the investigator. | Myocardial Infarction: ICD-9 DX: 410.xx ICD-10 DX: 110.xx, 122.xx ICD-10 DX: 121.xx, 122.xx Measured 180 days prior to and including the day of drug initiation in inpatient care setting, primary position: Heart Failure: ICD-9 DX: 428.xx, 398.91, 402.x1, 404.x1, 404.x3 ICD-10 DX: 109.81, 111.0, 113.0, 113.2, 150.xxx, 197.13x |
| | | NB. HF is included only if inpatient / primary position to detect the most severe cases as specified in the exclusion criterion of the trial |

| | | | 1 |
|---|---|---|---|
| | | Measured 180 days prior to and including the day of drug initiation: | |
| | | Anti-VEGFi CPT: 67028 (Intravitreal injection for pharmacologic agent) | |
| | | AND | |
| 7 | Proliferative retinopathy or maculopathy requiring acute treatment as judged by the investigator. | HCPCS: J9035 OR C9257 OR Q5107 (Bevacizumab 10 mg injection) OR<br>HCPCS: J2778 (Ranibizumab 0.1 mg) OR<br>HCPCS: C9291 OR Q2046 OR J0178 OR C9296 OR J9400 (Aflibercept 2 mg injection) | |
| | | Photocoagulation: CPT: 67228 (Panretinal photocoagulation) OR CPT: 67220 (Focal/Grid photocoagulation) OR CPT: 67028 (Intravitreal injection for pharmacologic agent) | |
| | | Measured 180 days prior to and including the day of drug initiation in any diagnosis position in the inpatient and outpatient and emergency care setting: | |
| | | Hypertensive crisis ICD-10 diagnosis: $116.x$ (includes hypertensive urgency, emergency, crisis, unspecified) | |
| | | OR | |
| 8 | Uncontrolled treated/untreated hypertension (systolic blood pressure ≥= 180 mmHg and/or diastolic blood pressure ≥= 100 mmHg). | Measured 180 days prior to and including the day of drug initiation in primary diagnosis position for inpatient or<br>any position for emergency care setting: | |
| | blood pressure >= 100 mmng). | Uncontrolled hypertension:<br>ICD-9 diagnosis: | |
| | | 401.9 (unspecified essential hypertension) 401.0 (malignant essential hypertension) | |
| | | 402.0x (malignant hypertensive heart disease) 403.0x (malignant hypertensive kidney disease) | |
| | | 404.0x (malignant hypertensive heart and kidney disease) 405.0x (malignant secondary hypertension) | |
| | | 403.9x (unspecified hypertensive kidney disease) 796.2 (elevated BP reading without Dx of HTN) | |
| | Cancer (except basal cell skin cancer or squamous cell skin cancer) or any clinically significant | Measured 1825 prior to and including the day of drug initiation in any diagnosis position and inpatient or outpatient care setting: | |
| 9 | Cancer (except basis cension cancer of squamous cension cancer) of any clinically significant disease or disorder, except for conditions associated to type 2 diabetes, which in the investigator's opinion could interfere with the results of the trial. | <u>Cancer:</u> | |
| | arrowgant of opinion could metrore with the regard of the filler. | ICD 9 diagnosis: 140.x-209.x (except 173.x, non-melanoma skin cancer and 209.4x, 209.5x, 209.6x) ICD 10 diagnosis: C00.x-C96, D45 (except C44.x, non-melanoma skin cancer) | |
| | | At least two measurements in the 180 days prior to and including the day of drug initiation inpatient or emergency department settings: | |
| 10 | Recurrent major hypoglycaemia as judged by the investigator. | Hypoglycemia: ICD-9 diagnosis: 251.0, 251.1, 251.2, 962.3, or 270.3 (primary position) or 250.8 without co-existence of 259.8, 272.7, | |
| | | 681.x,682.x, 686.9, 707.1–707.9, 730.0–730.2, or 731.8 (any position) ICD-10 diagnosis: E10.641, E11.641, E13.641, E10.649, E11.649, E13.649, E16.0, E16.1, E16.2 (primary position) or E11.69, E13.69, E10.69 without coexistence of E34.1, E34.8, E35, E75.2, E75.3, E77, L01, L02, L03, L97, M86, M90 | |
| N/A | Known or suspected allergy to trial product(s) or related products. | N/A | |
| | | Measured 90 days prior to and including the day of drug initiation: | |
| | | Injectable (IV) or (IM); | |
| 11 | Use of any drug (except for OADs), which in the investigator's opinion could interfere with glucose levels (e.g. systemic corticosteroids). | NDC Generic Name: methylprednisolone, hydrocortisone, dexamethasone CPT/HCPCS Procedure Code: J1020, J1030, J1040, J1720, J2920, J2930 | |
| | | Oral: | |
| | | NDC Generic Name: Cortisone, hydrocortisone, prednisone, prednisolone, methylprednisolone, dexamethasone | |
| N/A | Receipt of any investigational drug within the four weeks prior to this trial. | N/A | |
| N/A | Previous participation in the randomised phase of this trial. Re-screening is allowed once within the recruitment period. | N/A | |
| 14/24 | · | | |

| | | Manual 180 days single and including the day of days intrinsic in any dispersion of the contract of the contra | 1 |
|---|---|---|---|
| | | Measured 180 days prior to and including the day of drug initiation in any diagnosis position in inpatient or outpatient care setting: | |
| 12 | Known or suspected abuse of alcohol or narcotics. | Alcohol Abuse or Dependence ICD-9 diagnosis: 291.x, 303.xx, 305.9x, 357.5, 425.5, 535.30, 535.31, 571.0 - 571.3, 760.71, 790.3, 980.0, E860.0, E860.1, E860.8, E860.9, V11.3, V79.1 ICD-10 diagnosis: E24.4, F10.1xx (excluding F10.13x), F10.2xx, F10.9xx (excluding F10.93x), G31.2, G62.1, G72.1, 142.6, K29.2x, K70.xx, K85.2x, K86.0, O35.4, P04.3, Q86.0, R78.0, T51.0X1x, Z50.2, Z71.4, Z72.1 | |
| | | OR | |
| | | Drug Abuse or Dependence ICD-9 diagnosis: 292.xx, 304.xx, 305.xx (excluding 305.0x and 305.1), 648.3x, 779.5, 965.0x, 967.x, 969.xx, 970.xx, V65.42 ICD-10 diagnosis: F11.xxx, F12.xxx, F13.xxx, F14.xxx, F15.xxx, F16.xxx, F18.xxx, F19.xxx, O99.32x, P96.1, | |
| | | T40 mmm (amaladina T40 mm(n), T42 mmm (amaladina T42 mm(n), 771 51 | |
| | | Measured 180 days prior to and including the day of drug initiation in any diagnosis position in inpatient or outpatient care setting: | |
| 13 | Mental incapacity, unwillingness or language barrier precluding adequate understanding or cooperation. | Dementia and brain damages: ICD-9 diagnosis: 290.x, 294.x, 330.x, 331.x ICD-10 diagnosis: F01.50, F01.51, F02.80, F02.81, F03.90, F03.91, F04, F05, F06.x, F84.2, G13.2, G13.8, G30.x, G31.x, G91.x, G93.x, G94, E750, E751, E752, E754 NDC generic names: RIVASTIGMINE, DONEPEZIL HCL, ERGOLOID MESYLATES, GALANTAMINE HBR, MEMANTINE HCL, MEMANTINE HCL/DONEPEZIL HCL, RIVASTIGMINE TARTRATE, TACRINE HCL | |
| | | OR | |
| | | Non-compliance: ICD-9 diagnosis: V45-12, V15-81 | |
| 14 | Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures as | Measured 180 days prior to and including the day of drug initiation in any diagnosis position and inpatient or outpatient care setting: | |
| 14 | required by local law or practice). This exclusion criterion has been modified in Germany according to Substantial Protocol Amendment No. 2-DE, see Section 9.8.1. | Please refer to "Pregnancy definition" | |
| | | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: | |
| | | Contraindications to Glimepiride: | |
| | | Tyne 1 diabetes:<br>ICD 9 diagnosis: 250.01, 250.03, 250.11, 250.13, 250.21, 250.23, 250.31, 250.33, 250.41, 250.43, 250.51, 250.53, 250.61, 250.63, 250.71, 250.73, 250.81, 250.83, 250.91, 250.93<br>ICD 10 diagnosis: E10.x | |
| 15 | Any contraindications to metformin or glimepiride (according to local requirements). | Diabetic ketoacidosis (DKA):<br>ICD9 diagnosis: 250.1x<br>ICD10 diagnosis: E10.1x, E11.1x, E13.1x, E08.1x, E09.1x | |
| | | Other metabolic acidosis: ICD9 diagnosis: 276.2 ICD10 diagnosis: E87.2 | |
| 1 | | NB. All patients no treated with metformin at cohort entry have been excluded from the eligible cohort, assuming that all | |
| | | Measured 1825 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: | |
| 16 | Subjects with medical history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma (FMTC) if total thyroidectomy has not been performed or cannot be ensured (i.e. posterior capsule of the thyroid gland not removed). This exclusion criterion has been added only in | ICD-9 diagnosis: 258.02, 258.03<br>ICD-10 diagnosis: E31.22, E31.23 | |
| | Germany according to Substantial Protocol Amendment No. 2-DE, see Section 9.8.1. | NB. Thyroid carcinoma is already excluded with exclusion criterion 9 | |
| <u></u> | | 1 | |

| | PREGNANCY DEFINITION |
|---|---|
| 1. Delivery Codes | |
| Procedure Codes | Description |
| CPT-4 codes | |
| 1960 | Anesthesia for vaginal delivery only |
| 1961 | Anesthesia for cesarean delivery only |
| 1962 | Anesthesia for urgent hysterectomy following delivery |
| 1963 | Anesthesia for cesarean hysterectomy w/o any labor analgesia/anesthesia care |
| 1967 | Neuraxial labor analgesia/anesthesia, planned vaginal delivery |
| 1968 | Anesthesia for cesarean delivery following neuraxial labor analgesia/anesthesia |
| 1969 | Anes for cesarean hysterectomy following neuraxial labor analgesia/anesthesia |
| 59050 | Fetal monitoring in labor, physician w/written report; s & i |
| 59051 | Fetal monitoring in labor, physician w/written report; intrepretation only |
| 59400 | ROUTINE TOTAL OBSTETRIC CARE including antepartum care, vaginal delivery (with or without episiotomy, and/or forceps) and postpartum care. |
| 59409 | Vaginal delivery only (w/wo episiotomy &/or forceps) |
| 59410 | Vaginal delivery only (w/wo episiotomy &/or forceps); w/postpartum care |
| 59412 | Ext cephalic version, w/wo tocolysis |
| 59414 | Delivery of placenta (separate proc) |
| 59430 | Postpartum care only |
| 59510 | Routine obstetric care w/antepartum care, cesarean delivery, & postpartum care |
| 59514 | Cesarean delivery only |
| 59515 | Cesarean delivery only; w/postpartum care |
| 59525 | Subtotal/total hysterectomy after cesarean delivery |
| 59610 | Routine obstetric care including antepartum care, vaginal delivery (with or without episiotomy, and/or forceps) and postpartum care, after previous cesarean delivery |
| 59612 | Vaginal delivery only, after previous cesarean delivery (with or without episiotomy and/or forceps) |
| 59614 | Vaginal delivery only, previous cesarean delivery w/postpartum care |
| 59618 | Routine obstetric care including antepartum care, cesarean delivery, and postpartum care, following attempted vaginal delivery after previous cesarean delivery |
| 59620 | Cesarean delivery after failed vaginal delivery, previous cesarean delivery |
| 59622 | Cesarean delivery after failed vaginal delivery, previous cesarean delivery; w/postpartum care |
| 99436 | Attendance at delivery, at request of delivering physician, & stabilization of newborn |
| 99440 | Newborn resuscitation |
| ICD-9 procedure codes | |
| 72.xx | Forceps, vacuum, & breech |
| 73.xx | Other including manual delivery |
| 74xx | Cesarean section |
| 75.4x | Manual removal of placenta |
| ICD-10 procedure codes | |
| Normal Delivery | |
| 10E0XZZ | Delivery of Products of Conception, External Approach |
| C-Section | |
| 10D00Z0 | Extraction of Products of Conception, High, Open Approach |
| 10D00Z1 | Extraction of Products of Conception, Low, Open Approach |
| 10D00Z2 | Extraction of Products of Conception, Extraperitoneal, Open Approach |
| Other assisted delivery (fo | rceps, vacuum, internal version, other) |
| 10D07Z3 | Extraction of Products of Conception, Low Forceps, Via Natural or Artificial Opening |
| 10D07Z4 | Extraction of Products of Conception, Mid Forceps, Via Natural or Artificial Opening |
| 10D07Z5 | Extraction of Products of Conception, High Forceps, Via Natural or Artificial Opening |
| 10D07Z6 | Extraction of Products of Conception, Vacuum, Via Natural or Artificial Opening |
| 10D07Z7 | Extraction of Products of Conception, Internal Version, Via Natural or Artificial Opening |
| 10D07Z8 | Extraction of Products of Conception, Other, Via Natural or Artificial Opening |

#### 2. Identify preterm births Codes that have a specific gestational age mentioned Definition ICD-9 code 765.21 Less than 24 completed weeks of gestation 765.22 24 completed weeks of gestation 765.23 25-26 completed weeks of gestation 765.24 27-28 completed weeks of gestation 765.25 29-30 completed weeks of gestation 765.26 31-32 completed weeks of gestation 765.27 33-34 completed weeks of gestation 765.28 35-36 completed weeks of gestation ICD-10 code Definition P07.21 Extreme immaturity of newborn, gestational age less than 23 completed weeks P07.22 Extreme immaturity of newborn, gestational age 23 completed weeks P07.23 Extreme immaturity of newborn, gestational age 24 completed weeks P07.24 Extreme immaturity of newborn, gestational age 25 completed weeks P07.25 Extreme immaturity of newborn, gestational age 26 completed weeks P07.26 Extreme immaturity of newborn, gestational age 27 completed weeks P07.31 Preterm newborn, gestational age 28 completed weeks P07.32 Preterm newborn, gestational age 29 completed weeks P07.33 Preterm newborn, gestational age 30 completed weeks P07.34 Preterm newborn, gestational age 31 completed weeks P07.35 Preterm newborn, gestational age 32 completed weeks P07.36 Preterm newborn, gestational age 33 completed weeks P07.37 Preterm newborn, gestational age 34 completed weeks P07.38 Preterm newborn, gestational age 35 completed weeks P07.39 Preterm newborn, gestational age 36 completed weeks b. Codes indicating extreme prematurity ICD-9 code Definition 765 Disorders relating to extreme immaturity of infant 765.00 Extreme immaturity, unspecified [weight] 765.01 Extreme immaturity, less than 500 grams 765.02 Extreme immaturity, 500-749 grams 765.03 Extreme immaturity, 750-999 grams 765.04 Extreme immaturity, 1,000-1,249 grams 765.05 Extreme immaturity, 1,250-1,499 grams 765.06 Extreme immaturity, 1,500-1,749 grams 765.07 Extreme immaturity, 1,750-1,999 grams 765.08 Extreme immaturity, 2,000-2,499 grams ICD-10 code Definition P07.2 Extreme immaturity of newborn P07.20 Extreme immaturity of newborn, unspecified weeks of gestation 042.012 Preterm premature rupture of membranes, onset of labor within 24 hours of rupture, second trimester c. Other preterm codes Definition ICD-9 code 765.1 Disorders relating to other preterm infants 765.10 Other preterm infants, unspecified [weight] Other preterm infants, less than 500 grams 765.11 765.12 Other preterm infants, 500-749 grams 765.13 Other preterm infants, 750-999 grams

| 765.14 | Other preterm infants, 1,000-1,249 grams |
|---|---|
| 765.15 | Other preterm infants, 1,250-1,499 grams |
| 765.16 | |
| | Other preterm infants, 1,500-1,749 grams |
| 765.17 | Other preterm infants, 1,750-1,999 grams |
| 765.18 | Other preterm infants, 2,000-2,499 grams |
| 644.21 | Onset of delivery before 37 completed weeks of gestation |
| ICD-10 code | Definition 500 hours of the state of the sta |
| P05.01 | Disorders of newborn related to slow fetal growth and fetal malnutrition less than 500 grams |
| P05.02 | Disorders of newborn related to slow fetal growth and fetal malnutrition, 500-749 grams |
| P05.03 | Disorders of newborn related to slow fetal growth and fetal malnutrition, 750-999 grams |
| P05.04 | Disorders of newborn related to slow fetal growth and fetal malnutrition, 1000-1249 grams |
| P05.05 | Disorders of newborn related to slow fetal growth and fetal malnutrition, 1250-1499 grams |
| P05.06 | Disorders of newborn related to slow fetal growth and fetal malnutrition, 1500-1749 grams |
| P05.11 | Newborn small for gestational age, less than 500 grams |
| P05.12 | Newborn small for gestational age, 500-749 grams |
| P05.13 | Newborn small for gestational age, 750-999 grams |
| P05.14 | Newborn small for gestational age, 1000-1249 grams |
| P05.15 | Newborn small for gestational age, 1250-1499 grams |
| P05.16 | Newborn small for gestational age, 1500-1749 grams |
| P07.01 | Extremely low birth weight newborn, less than 500 grams |
| P07.02 | Extremely low birth weight newborn, 500-749 grams |
| P07.03 | Extremely low birth weight newborn, 750-999 grams |
| P07.14 | Other low birth weight newborn,1000-1249 grams |
| P07.15 | Other low birth weight newborn,1250-1499 grams |
| P07.16 | Other low birth weight newborn, 1500-1749 grams |
| P07.3 | Preterm [premature] newborn [other] |
| P07.30 | Preterm newborn, unspecified weeks of gestation |
| 060.1 | Preterm labor with preterm delivery |
| 042.01 | Preterm premature rupture of membranes, onset of labor within 24 hours of rupture |
| 042.019 | Preterm premature rupture of membranes, onset of labor within 24 hours of rupture, unspecified trimester |
| 042.013 | Preterm premature rupture of membranes, onset of labor within 24 hours of rupture, third trimester |
| Other Codes | Description |
| ICD-9 | |
| 644.2 | early onset of delivery |
| 644.2 | Early onset of delivery, unspecified as to episode of care or not applicable |
| 644.21 | Early onset of delivery, delivered, with or without mention of antepartum condition |
| 776.6 | anemia of prematurity |
| 362.2 | retinopathy of prematurity, unspecified |
| 362.22 | retinopathy of prematurity, stage 0 |
| 362.23 | retinopathy of prematurity, stage 1 |
| 362.24 | retinopathy of prematurity, stage 2 |
| 362.25 | retinopathy of prematurity, stage 3 |
| 362.26 | retinopathy of prematurity, stage 4 |
| 362.27 | retinopathy of prematurity, stage 5 |
| CPT | Technopathy or prematerity, stage of |
| 49491 | repair, initial inguinal hernia, preterm infant (younger than 37 weeks gestation at birth), performed from birth up to 50 weeks postconception |
| 49492 | repair, initial inguinal hernia, preterm infant (younger than 37 weeks gestation at birth), performed from birth up to 50 weeks postconception |
| 67229 | treatment of extensive or progressive retinopathy, 1 or more sessions; preterm infant (less than 37 weeks gestation at birth), performed from |
| 836 | anesthesia for hernia repairs in the lower abdomen not otherwise specified, infants younger than 37 weeks gestational age at birth |
| ICD-10 code | Definition |

| H35.1 | Retinopathy of prematurity |
|---|---|
| P61.2 | Anemia of prematurity |
| | V for ICD-9 and Z for ICD-10 codes excluded) |
| ICD9 Code | Description |
| V27.2 | Twins both liveborn |
| V27.3 | Mother with twins one liveborn and one stillborn |
| V27.4 | Mother with twins both stillborn |
| V27.5 | Other multiple birth, all liveborn |
| V27.6 | Other multiple birth, some liveborn |
| V31 | Twin, mate liveborn |
| V32 | Twin birth mate stillborn |
| V33 | Twin, unspecified |
| V34 | Other multiple, mates all liveborn |
| V35 | Other multiple birth (three or more) mates all stillborn |
| V36 | Other multiple, mates live- and stillborn |
| V37 | Other multiple, unspecified |
| 651 | Multiple gestation |
| 651.0x | Twin Pregnancy |
| 651.1x | Triplet pregnancy |
| 651.2x | Quadruplet pregnancy |
| 651.3x | Twin pregnancy with fetal loss and retention of one fetus |
| 651.4x | Triplet pregnancy with fetal loss and retention of one or more fetus(es) |
| 651.5x | Quadruplet pregnancy with fetal loss and retention of one or more fetus(es) |
| 651.6x | Other multiple pregnancy with fetal loss and retention of one or more fetus(es) |
| 651.7x | Multiple gestation following (elective) fetal reduction |
| 651.8x | Other specified multiple gestation |
| 651.9x | Unspecified multiple gestation |
| 652.6x | Multiple gestation with malpresentation of one fetus or more |
| 660.5x | Locked Twins |
| 662.3x | Delayed delivery of second twin, triplet, etc. |
| 761.5x | Multiple pregnancy |
| ICD10 Code | Description |
| O30xxxx | Multiple gestation |
| O31xxxx | Complications specific to multiple gestation |
| 043.02 | Fetus-to-fetus placental transfusion syndrome |
| 063.2 | Delayed delivery of second twin, triplet, etc. |
| Z37.2 | Twins, both liveborn |
| Z37.3 | Twins, one liveborn and one stillborn |
| Z37.5 | Other multiple births, all liveborn |
| Z37.50 | Multiple births, unspecified, all liveborn |
| Z37.51 | Triplets, all liveborn |
| Z37.52 | Quadruplets, all liveborn |
| Z37.53 | Quintuplets, all liveborn |
| Z37.54 | Sextuplets, all liveborn |
| Z37.59 | Other multiple births, all liveborn |
| Z37.6 | Other multiple births, some liveborn |
| Z37.60 | Multiple births, unspecified, some liveborn |
| Z37.61 | Triplets, some liveborn |
| Z37.62 | Quadruplets, some liveborn |
| Z37.63 | Quintuplets, some liveborn |

| Z37.64 | Sextuplets, some liveborn |
|---|---|
| Z37.69 | Other multiple births, some liveborn |
| Z38.3 | Twin liveborn infant, born in hospital |
| Z38.30 | Twin liveborn infant, delivered vaginally |
| Z38.31 | Twin liveborn infant, delivered by cesarean |
| Z38.4 | Twin liveborn infant, born outside hospital |
| Z38.5 | Twin liveborn infant, unspecified as to place of birth |
| Z38.6 | Other multiple liveborn infant, born in hospital |
| Z38.61 | Triplet liveborn infant, delivered vaginally |
| Z38.62 | Triplet liveborn infant, delivered by cesarean |
| Z38.63 | Quadruplet liveborn infant, delivered vaginally |
| Z38.64 | Quadruplet liveborn infant, delivered by cesarean |
| Z38.65 | Quintuplet liveborn infant, delivered vaginally |
| Z38.66 | Quintuplet liveborn infant, delivered by cesarean |
| Z38.68 | Other multiple liveborn infant, delivered vaginally |
| Z38.69 | Other multiple liveborn infant, delivered by cesarean |
| Z38.7 | Other multiple liveborn infant, born outside hospital |
| Z38.8 | Other multiple liveborn infant, unspecified as to place of birth |
| P01.5 | Newborn affected by multiple pregnancy |
| 3. Post-Term Code | 25 |
| ICD-9 code | Definition |
| 645 | Late Pregnancy |
| 645.1 | Post term pregnancy |
| 645.1 | Post term pregnancy, unspecified as to episode of care or not applicable |
| 645.11 | Post term pregnancy, delivered, with or without mention of antepartum condition |
| 645.13 | Post term pregnancy, antepartum condition or complication |
| 645.2 | Prolonged pregnancy |
| 645.2 | Prolonged pregnancy, unspecified as to episode of care or not applicable |
| 645.21 | Prolonged pregnancy, delivered, with or without mention of antepartum condition |
| 645.23 | Prolonged pregnancy, antepartum condition or complication |
| 766.2 | Late infant, not 'heavy-for-dates' |
| 766.21 | Post-term infant |
| 766.22 | Prolonged gestation of infant |

ICD-10 code Definition
O48 Late pregnancy
O48.0 Post-term pregnancy
O48.1 Prolonged pregnancy

P08.2 Late newborn, not heavy for gestational age

P08.21 Post-term newborn

P08.22 Prolonged gestation of newborn Z3A.41 41 weeks gestation of pregnancy Z3A.42 42 weeks gestation of pregnancy

Z3A.49 Greater than 42 weeks gestation of pregnancy

#### 4. Codes indicating a prenatal care visit:

ICD-9: V220x, V221x, V23xx

#### Anti-diabetic treatments (other than insulin)

### 1st and 2nd Generation Sus (excluding glimepiride)

GLIPIZIDE/METFORMIN HCL

**ACETOHEXAMIDE** 

GLYBURIDE, MICRONIZED

**TOLBUTAMIDE** 

GLYBURIDE/METFORMIN HCL

TOLAZAMIDE

**CHLORPROPAMIDE** 

**GLYBURIDE** 

**GLIPIZIDE** 

#### **AGIs**

**ACARBOSE** 

**MIGLITOL** 

#### **DPP-4 Inhibitors**

ALOGLIPTIN BENZOATE

DAPAGLIFLOZIN PROPANEDIOL/SAXAGLIPTIN HCL

ERTUGLIFLOZIN PIDOLATE/SITAGLIPTIN PHOSPHATE

SAXAGLIPTIN HCL/METFORMIN HCL

LINAGLIPTIN

ALOGLIPTIN BENZOATE/METFORMIN HCL

ALOGLIPTIN BENZOATE/PIOGLITAZONE HCL

EMPAGLIFLOZIN/LINAGLIPTIN

SAXAGLIPTIN HCL

SITAGLIPTIN PHOSPHATE/METFORMIN HCL

SITAGLIPTIN PHOSPHATE/SIMVASTATIN

SITAGLIPTIN PHOSPHATE

#### Glitazones

ALOGLIPTIN BENZOATE/PIOGLITAZONE HCL

PIOGLITAZONE HCL

PIOGLITAZONE HCL/GLIMEPIRIDE

PIOGLITAZONE HCL/METFORMIN HCL

ROSIGLITAZONE MALEATE

ROSIGLITAZONE MALEATE/GLIMEPIRIDE

ROSIGLITAZONE MALEATE/METFORMIN HCL

#### **GLP-1** RA (excluding liraglutide monotherapy)

ALBIGLUTIDE

DULAGLUTIDE

**EXENATIDE** 

**EXENATIDE MICROSPHERES** 

INSULIN DEGLUDEC/LIRAGLUTIDE

INSULIN GLARGINE, HUMAN RECOMBINANT ANALOG/LIXISENATIDE

LIXISENATIDE

**SEMAGLUTIDE** 

#### Meglitinides

**NATEGLINIDE** 

REPAGLINIDE

REPAGLINIDE/METFORMIN HCL

#### **SGLT-2 Inhibitors**

CANAGLIFLOZIN

CANAGLIFLOZIN/METFORMIN HCL

DAPAGLIFLOZIN PROPANEDIOL/SAXAGLIPTIN HCL

ERTUGLIFLOZIN PIDOLATE

ERTUGLIFLOZIN PIDOLATE/SITAGLIPTIN PHOSPHATE

DAPAGLIFLOZIN PROPANEDIOL/METFORMIN HCL

EMPAGLIFLOZIN/LINAGLIPTIN

**EMPAGLIFLOZIN** 

DAPAGLIFLOZIN PROPANEDIOL

ERTUGLIFLOZIN PIDOLATE/METFORMIN HCL

EMPAGLIFLOZIN/METFORMIN HCL

#### Insulin

#### **Bolus insulins**

**INSULIN GLULISINE** 

INSULIN REGULAR, BEEF-PORK

**INSULIN ASPART (NIACINAMIDE)** 

INSULIN REGULAR, HUMAN/INSULIN RELEASE UNIT

INSULIN REGULAR, HUMAN BUFFERED

INSULIN REGULAR, HUMAN/INSULIN RELEASE UNIT/CHAMBER/INHALER

**INSULIN ASPART** 

INSULIN ASPART PROTAMINE HUMAN/INSULIN ASPART

INSULIN LISPRO PROTAMINE AND INSULIN LISPRO

**INSULIN LISPRO** 

INSULIN REGULAR, HUMAN

**Intermediate and Long-acting Insulins** 

**INSULIN DEGLUDEC** 

**INSULIN DETEMIR** 

INSULIN DEGLUDEC/LIRAGLUTIDE

INSULIN NPH HUMAN AND INSULIN REGULAR HUMAN SEMI-SYNTHETIC

INSULIN NPH HUMAN SEMI-SYNTHETIC

INSULIN ISOPHANE NPH, BF-PK

INSULIN GLARGINE, HUMAN RECOMBINANT ANALOG/LIXISENATIDE

INSULIN GLARGINE, HUMAN RECOMBINANT ANALOG

INSULIN NPH HUMAN ISOPHANE

INSULIN NPH HUMAN ISOPHANE/INSULIN REGULAR, HUMAN

## Appendix B



## Appendix B

| <del>-</del> | | UNMATCHED | |
|---|---|---|---|
| | | Optum | |
| Variable<br>Number of patients | Glimpiride<br>3,096 | Liraglutide<br>378 | St. Diff |
| Age squared | | | |
| mean (sd) ge (continuous) | 761406 (223830.2) | 651214 (225218.8) | 0.491 |
| mean (sd)<br>te (categories) | 64.24 (10.37) | 59.22 (10.94) | 0.471 |
| 8 - 40; n (%) | 95 (3.1%) | 20 (5.3%) | -0.110 |
| 1 -50; n (%)<br>1 -60; n (%) | 266 (8.6%)<br>602 (19.4%) | 64 (16.9%)<br>106 (28.0%) | -0.251<br>-0.203 |
| - 70; n (%)<br>- 80; n (%) | 1187 (38.3%) | 133 (35.2%)<br>55 (14.6%) | 0.064<br>0.390 |
| ler | 946 (30.6%) | | |
| : MALE; n (%)<br>FEMALE; n (%) | 1726 (55.7%)<br>1370 (44.3%) | 179 (47.4%)<br>199 (52.6%) | 0.167<br>-0.167 |
| ite; n (%)<br>white; n (%) | 1492 (48.2%)<br>1604 (51.8%) | 220 (58.2%)<br>158 (41.8%) | -0.201<br>0.201 |
| ndar time years (Jan 2010 - Jun 2020) | | | |
| n 26, 2010 - Dec 31, 2017; n (%)<br>n 1, 2018 - Jun 30, 2020; n (%) | 1850 (59.8%)<br>1246 (40.2%) | 255 (67.5%)<br>123 (32.5%) | -0.161<br>0.161 |
| al Health | | | |
| ng; n (%)<br>y or Overweight; n (%) | 296 (9.6%)<br>760 (24.5%) | 30 (7.9%)<br>93 (24.6%) | 0.060<br>-0.002 |
| ty; n (%)<br>reight: n (%) | 554 (17.9%)<br>247 (8.0%) | 79 (20.9%)<br>16 (4.2%) | -0.076<br>0.159 |
| ned comorbidity score, 180 days | | | |
| (sd)<br>core: Empirical Version 180 days | 2.06 (1.56) | 1.86 (1.36) | 0.137 |
| (sd) | 0.99 (0.77) | 1.03 (0.73) | -0.053 |
| bA1c | 8.16 (0.96) | 8.18 (0.99) | -0.021 |
| sd)<br>scular Comorbidities | | | |
| sion; n (%)<br>demia; n (%) | 391 (12.6%)<br>2296 (74.2%) | 66 (17.5%)<br>299 (79.1%) | -0.137<br>-0.116 |
| erosis Disease (MI, angina, CAD and other forms of chronic ischemic | 566 (18.3%) | 43 (11.4%) | 0.116 |
| ease, History of CABG or PTCA); n (%)<br>: n (%) | 64 (2.1%) | 3 (0.8%) | 0.195 |
| vII; n (%) | 10 (0.3%) | 1 (0.3%) | 0.000 |
| nstable angina; n (%)<br>angina; n (%) | 18 (0.6%)<br>80 (2.6%) | 1 (0.3%)<br>6 (1.6%) | 0.045<br>0.070 |
| other forms of chronic ischemic heart disease; n (%) | 415 (13.4%) | 30 (7.9%) | 0.179 |
| y of CABG or PTCA; n (%) | 107 (3.5%) | 9 (2.4%) | 0.065 |
| r PAD surgery; n (%)<br>vascular disease (Stroke, TIA, Late effects); n (%) | 166 (5.4%)<br>77 (2.5%) | 11 (2.9%)<br>2 (0.5%) | 0.126<br>0.165 |
| e (Ischemic or hemorrhagic); n (%) | 40 (1.3%) | 1 (0.3%) | 0.112 |
| n (%)<br>effects of cerebrovascular disease; n (%) | 27 (0.9%)<br>28 (0.9%) | 1 (0.3%)<br>0 (0.0%) | 0.078<br>0.135 |
| ailure; n (%)<br>brillation: n (%) | 103 (3.3%) | 10 (2.6%) | 0.041 |
| illation; n (%)<br>diac dysrhythmia; n (%) | 121 (3.9%)<br>190 (6.1%) | 14 (3.7%)<br>18 (4.8%) | 0.010<br>0.057 |
| s Mellitus Comorbidities | | | |
| remia; n (%)<br>nephropathy; n (%) | 20 (0.6%)<br>434 (14.0%) | 4 (1.1%)<br>48 (12.7%) | -0.054<br>0.038 |
| Neuropathy; n (%) | 495 (16.0%) | 60 (15.9%) | 0.003 |
| : Retinopathy; n (%)<br>is with unspecified complications; n (%) | 134 (4.3%)<br>122 (3.9%) | 20 (5.3%)<br>14 (3.7%) | -0.047<br>0.010 |
| es with peripheral circulatory disorders and amputations, DF; n (%)* | 70 (2.3%) | 9 (2.4%) | -0.007 |
| etes with peripheral circulatory disorders; n (%)<br>er-limb amputations; n (%) | 38 (1.2%)<br>4 (0.1%) | 5 (1.3%)<br>1 (0.3%) | -0.009<br>-0.045 |
| tic Foot; n (%) | 32 (1.0%) | 3 (0.8%) | 0.021 |
| omorbidities<br>: kidney disease stages I-IV and NOS; n (%) | 381 (12.3%) | 40 (10.6%) | 0.053 |
| laneous renal disease; n (%) | 109 (3.5%) | 10 (2.6%) | 0.052 |
| disorders (Anxiety and Depression); n (%)<br>ety; n (%) | 332 (10.7%)<br>211 (6.8%) | 47 (12.4%)<br>27 (7.1%) | -0.053<br>-0.012 |
| sion; n (%) | 162 (5.2%) | 28 (7.4%) | -0.091 |
| morbidities<br>ive sleep apnea; n (%) | 259 (8.4%) | 41 (10.8%) | -0.082 |
| %) | 207 (6.7%) | 9 (2.4%) | 0.207 |
| n (%)<br>hrosis: n (%) | 96 (3.1%)<br>363 (11.7%) | 14 (3.7%)<br>49 (13.0%) | -0.033<br>-0.040 |
| FLD; n (%) | 98 (3.2%) | 16 (4.2%) | -0.053 |
| ons | 2585 (83.5%) | 324 (85.7%) | -0.061 |
| rtensive medications; n (%)<br>RBs; n (%) | 2257 (72.9%) | 285 (75.4%) | -0.061 |
| ckers; n (%)<br>channel blockers; n (%) | 971 (31.4%)<br>795 (25.7%) | 94 (24.9%)<br>83 (22.0%) | 0.145<br>0.087 |
| channel blockers; n (%)<br>: n (%) | 369 (11.9%) | 52 (13.8%) | -0.057 |
| cs; n (%) | 1108 (35.8%) | 133 (35.2%) | 0.013 |
| ther lipid-lowering drugs; n (%)<br>: n (%) | 2402 (77.6%)<br>2285 (73.8%) | 291 (77.0%)<br>273 (72.2%) | 0.014<br>0.036 |
| (%) | 370 (12.0%) | 49 (13.0%) | -0.030 |
| zing Medications; n (%) | 507 (16.4%)<br>719 (23.2%) | 72 (19.0%)<br>129 (34.1%) | -0.068<br>-0.243 |
| ts; n (%) | 540 (17.4%) | 105 (27.8%) | -0.251 |
| /hypnotics; n (%)<br>pine; n (%) | 114 (3.7%)<br>256 (8.3%) | 25 (6.6%)<br>42 (11.1%) | -0.131<br>-0.095 |
| ids; n (%) | 319 (10.3%) | 49 (13.0%) | -0.084 |
| lization<br>dication claims | | | |
| 1) | 11.47 (6.60) | 12.82 (6.94) | -0.199 |
| of office visits<br>sd) | 4.76 (3.58) | 5.24 (3.72) | -0.131 |
| hospitalizations or ED visits | | | |
| )<br>Endocrinologist visits | 0.24 (0.87) | 0.20 (0.66) | 0.052 |
| sd) | 0.13 (0.55) | 0.27 (0.85) | -0.196 |
| of HbA1c test orders<br>sd) | 1.77 (0.68) | 1.79 (0.78) | -0.012 |
| i)<br>lexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy (CRC | 1.77 (0.68) | 1.79 (0.78) | -0.012 |
| ng); n (%) | | ,, | |
| | 400 (12.9%)<br>120 (3.9%) | 59 (15.6%)<br>16 (4.2%) | -0.077<br>-0.015 |
| | 659 (21.3%) | 93 (24.6%) | -0.079 |
| r of Pap smear (Cervical cancer screening); n (%)<br>cine; n (%) | 671 (21.7%) | 82 (21.7%) | 0.000 |
| of Pap smear (Cervical cancer screening); n (%) ine; n (%) scoccal vaccine; n (%) | | 0.03 (0.18) | 0.002 |
| r of Paps smear (Cervical cancer screening); n (%) icine; n (%) scoccal vaccine; n (%) or DDXA tests (sd) | 0.04 (0.19) | 0.03 (0.18) | |
| of Paps mear (Cervical cancer screening); n (%) ine; n (%) occacial vaccine; n (%) of DXA tests (sd) or pharmacy cost (charges in U.S. \$) | | | -D 331 |
| of Pap smear (Cervical cancer screening); n (%) ne, n (%) occcal waccine; n (%) of DXA tests (sd) pn pharmacy cost (charges in U.S. \$) (sd) (st) | 180.68 (259.85) | 280.36 (336.80) | -0.331 |
| r of Pags maser (Cervical cancer screening); n (%) cinen; n(%) occoccal vaccine; n (%) or of DXA Nestes (s)dH (s)dH (s)dH (s)dSH | 180.68 (259.85)<br>1016 (32.8%) | 280.36 (336.80) | -0.421 |
| per of Mammograms (Breast cancer screening); n (%) ere of Pay smear (Evrival cancer screening); n (%) ccine, n (%) ere of Pay shear (Evrival cancer screening); n (%) ere of DXA tests in (d) y for pharmacy cost (charges in U.S. 5) in (d) est type emmercal; n (%) intercal; n (%) illicare, n (%) illicare, n (%) illicare, n (%) illicare, n (%) | 180.68 (259.85)<br>1016 (32.8%)<br>2080 (67.2%) | 280.36 (336.80)<br>201 (53.2%)<br>177 (46.8%) | -0.421<br>0.421 |
| re of Pap smear (Cervical cancer screening); n (%) cincen (%) nococcal vasccinen (%) n (sd) for pharmacy cost (charges in U.S. 5) n (sd) for pharmacy cost (charges in U.S. 5) set type mecial; n (%) (cincen (%) cilcen (%) (cilcen (%) (cilcen (%) (cilcen (%) (cilcen (%)) | 180.68 (259.85)<br>1016 (32.8%) | 280.36 (336.80) | -0.421 |
| re of Pap smee (Cervical cancer screening); n (%) (inen, 16%) conceal waccine, n (%) conceal waccine, n (%) contact waccine, n (%) (bd) (br) (br) (br) (br) (br) (br) (br) (br | 180.68 (259.85)<br>1016 (32.8%)<br>2080 (67.2%) | 280.36 (336.80)<br>201 (53.2%)<br>177 (46.8%) | -0.421<br>0.421 |

<sup>\*</sup> variables included in the PS model # copay of index drugs is not included